CLINICAL TRIAL: NCT04132752
Title: Does Motivation of the Parents Affect the Efficiency of Home Exercises in Children With OBPP?
Brief Title: Motivation's Effect on Home Exercise in Children With OBPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tüzün Fırat, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HacettepeOBPPhome
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Obstetric Paralyses
Keywords: obstetric paralysis; home exercise; motivation; rehabilitation; parents
MeSH Terms: conditions — Paralysis, Obstetric | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Intervention Model Description: 33 children with obstetric brachial plexus palsy (OBPP) were randomized into control or intervention groups. Both groups parents were informed about OBPP, given home exercise and exercise diary. Intervention group was called via phone weekly in order to motivate and answer questions. Children's functional scores and parents motivation was measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents were informed about obstetric brachial plexus palsy, given home exercise program and exercise diary.
  Interventions: Other: Motivation
- Control (No Intervention): Parents were informed about obstetric brachial plexus palsy, given home exercise program and exercise diary.

INTERVENTIONS:
Other: Motivation — Families were called via phone weekly and all questions were answered. Parents were motivated through phone.
  Arms: Intervention

SUMMARY:
The present study examined the effect of motivation on home exercise program and children's functional scores. 33 OBPP children (Narakas Type 2) aged between 0-18 months were divided into two groups. Intervention group was motivated via phone. Both groups were informed about OBPP, performed home exercises and filled exercise diary. Intrinsic Motivation Scale was used for measuring motivation and Gilbert and Raimondi Scoring and Active Movement Scoring were used for evaluating functional improvements at first assessment, 6th week and 12th week. For final comparison, parents were divided into two more groups (highly motivated and motivated group) based on motivation scores.

DETAILED DESCRIPTION:
Home exercise program is widely used for treatment of OBPP children. The present study examined the effect of motivation on home exercise program and children's functional scores. 33 OBPP children (Narakas Type 2) aged between 0-18 months were divided into two groups. Intervention group was motivated via phone. Both groups were informed about OBPP, performed home exercises and filled exercise diary. Intrinsic Motivation Scale was used for measuring motivation and Gilbert and Raimondi Scoring and Active Movement Scoring were used for evaluating functional improvements at first assessment, 6th week and 12th week. For final comparison, parents were divided into two more groups (highly motivated and motivated group) based on motivation scores.

ELIGIBILITY:
Inclusion Criteria:

* Being classified as Narakas type 2a or 2b
* Being aged between 0 - 18 months
* Not having regular physiotherapy and rehabilitation program

Exclusion Criteria:

* Having a clinical condition such as upper motor neuron lesion that may affect child's affected arm or whole body,
* Having secondary surgery for orthopedic problems within last 6 months.
* Mother having an unidentified cognitive problem,
* Parents having another child with a disability,
* Parents not willing to participate.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Motivation change | From baseline to 12th week
  Intrinsic motivation scale measurement: has 21 questions with likert scale rating 1 to 7. Lowest score 21; meaning not motivated at all, 84 means neutral and 147 means fully motivated.
Scoring general arm function | From baseline to 12th week
  Active Movement Scale was used for scoring arm function: scale is scored from 1 to 5, with 1 being the worst and 5 being best functional status.
Scoring shoulder function | From baseline to 12th week
  Gilbert and Raimondi's scale was used for scoring shoulder function: scale is scored from 1 to 5, with 1 being the worst and 5 being best functional status.

SECONDARY OUTCOMES:
Scoring elbow function | From baseline to 12th week
  Gilbert scale was used for scoring elbow function: scale is scored from 1 to 5, with 1 being the worst and 5 being best functional status.
Scoring hand function | From baseline to 12th week
  Raimondi's scale was used for scoring hand function: scale is scored from 1 to 5, with 1 being the worst and 5 being best functional status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtis C, Stephens D, Clarke HM, Andrews D. The active movement scale: an evaluative tool for infants with obstetrical brachial plexus palsy. J Hand Surg Am. 2002 May;27(3):470-8. doi: 10.1053/jhsu.2002.32965. PMID 12015722
- [Background] James MA. Use of the Medical Research Council muscle strength grading system in the upper extremity. J Hand Surg Am. 2007 Feb;32(2):154-6. doi: 10.1016/j.jhsa.2006.11.008. No abstract available. PMID 17275587
- [Background] Nijenhuis SM, Prange GB, Amirabdollahian F, Sale P, Infarinato F, Nasr N, Mountain G, Hermens HJ, Stienen AH, Buurke JH, Rietman JS. Feasibility study into self-administered training at home using an arm and hand device with motivational gaming environment in chronic stroke. J Neuroeng Rehabil. 2015 Oct 9;12:89. doi: 10.1186/s12984-015-0080-y. PMID 26452749
- [Background] Bialocerkowski A, Kurlowicz K, Vladusic S, Grimmer K. Effectiveness of primary conservative management for infants with obstetric brachial plexus palsy. Int J Evid Based Healthc. 2005 Mar;3(2):27-44. doi: 10.1111/j.1479-6988.2005.00020.x. PMID 21631743